CLINICAL TRIAL: NCT03320135
Title: Enamel Matriz Derivate for Treatment of Proximal Class II Furcation Defects: a Randomized Clinical Trial
Brief Title: EMD for Treatment of Proximal Class-II Furcation Involvements
Acronym: OFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, DDS,MS,PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF ICT
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Generalized Aggressive Periodontitis
Keywords: enamel matrix derivative; proximal furcation; randomized clinical trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enamel matrix derivative proteins (Active Comparator): Open flap debridement to enamel matrix derivative application in proximal class-II furcation.
  Interventions: Procedure: Enamel matrix derivative proteins; Procedure: Open Flap debridement
- Open Flap Debridement (Active Comparator): Open flap debridement in proximal class-II furcation.
  Interventions: Procedure: Open Flap debridement

INTERVENTIONS:
Procedure: Enamel matrix derivative proteins — Open flap debridement to enamel matrix derivative to treat proximal furcation involvements.
  Other Names: Surgical therapy
  Arms: Enamel matrix derivative proteins
Procedure: Open Flap debridement — Open flap debridement will be performed to decontaminate the proximal furcation involvements.
  Other Names: Surgical therapy

SUMMARY:
The aim of the present study is to evaluate the clinical response of proximal furcations treated with enamel matrix derivative proteins (EMD).

DETAILED DESCRIPTION:
Proximal class-II furcation represents a challeng to periodontal therapy. Studies show that the ultrasonic non-surgical therapy doesn't work in these defects and the guided tissue regeneration therapy with membranes also demonstrates an unpredictable improvement. Therefore, enamel matrix derivative proteins (EMD) have been proposed as a periodontal regenerative procedure due to their fundamental role in cementum development.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized aggressive periodontitis (Armitage, 1999; American Academy of Periodontology, 2015);
* Have undergone a first approach for periodontal treatment (full-mouth ultrasonic debridement);
* Presence of one proximal class-II furcation presenting probing depth > 4 mm and bleeding on probing ;
* Good general health;
* Agree to participate in the study and sign the informed consent form (TCLE) after explaining the risks and benefits;

Exclusion Criteria:

* Systemic problems (cardiovascular alterations, blood dyscrasias, immunodeficiency - ASA III / IV / V) that contraindicate the periodontal procedure;
* Have used antibiotics and anti-inflammatories in the last six months;
* Smoke ≥ 10 cigarettes/day;
* Pregnant or lactating;
* Chronic use of medications that may alter the response of periodontal tissues;
* Indication of antibiotic prophylaxis for dental procedures;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Horizontal clinical attachment level | 1 year
  horizontal component of the defect

CONTACTS AND LOCATIONS:
Overall Officials: Mauro M Santamaria, DDS, PhD, Study Director — Universidade Estadual Paulista "Julio de Mesquita Filho", ICT/UNESP
Locations (1):
- Naira Andere, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Result] Casarin RC, Del Peloso Ribeiro E, Nociti FH Jr, Sallum AW, Sallum EA, Ambrosano GM, Casati MZ. A double-blind randomized clinical evaluation of enamel matrix derivative proteins for the treatment of proximal class-II furcation involvements. J Clin Periodontol. 2008 May;35(5):429-37. doi: 10.1111/j.1600-051X.2008.01202.x. Epub 2008 Mar 12. PMID 18341602